CLINICAL TRIAL: NCT07255794
Title: Comparison of the Effects of Dynamic Neuromuscular Stabilization and Thoracic Stabilization Exercises on Thoracic Erector Spinae Muscle Strength Using EMG Biofeedback in Individuals With Kyphosis
Brief Title: DNS vs Thoracic Stabilization Exercises in Thoracic Kyphosis
Acronym: TK-DNS-TS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esra BECENI (Other)
Responsible Party: Sponsor-Investigator, Esra BECENI, lecturer, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-FHP-DNS-TS-2025-02
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Kyphosis
Keywords: dynamic neuromuscular stabilization(DNS); electromyography; thoracic stabilization exercises
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Intervention Model Description: a randomized, controlled, assessor-blind, prospective study
Who Masked: Outcomes Assessor
Masking Description: Randomization will be done by the sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Neuromuscular Stabilization (DNS) Group (DNSG) (Experimental)
  Interventions: Behavioral: Dynamic Neuromuscular Stabilization Exercises
- Thoracic Stabilization Exercise Group (TSG) (Experimental)
  Interventions: Behavioral: Thoracic Stabilization Exercise

INTERVENTIONS:
Behavioral: Dynamic Neuromuscular Stabilization Exercises — Participants in the DNS group will perform Dynamic Neuromuscular Stabilization exercises based on developmental kinesiology. The program includes prone (4.5-month position), modified prone over a Swiss ball, quadruped (9-month position) and prone exercises on a Swiss ball with bilateral hand support. All exercises emphasize proper spinal alignment, diaphragmatic breathing and coordinated activation of the deep stabilizing muscles. Participants will complete two supervised sessions per week and perform home exercises twice daily (10 repetitions per exercise) for 6 weeks. An exercise diary will be used to monitor adherence.
  Arms: Dynamic Neuromuscular Stabilization (DNS) Group (DNSG)
Behavioral: Thoracic Stabilization Exercise — Participants in the thoracic stabilization group will perform a structured thoracic and scapular stabilization program including foam roller thoracic extension in supine, prone thoracic extension, child's pose with thoracic extension and scapular retraction exercises. The exercises are designed to improve thoracic mobility, strengthen the thoracic extensors and enhance postural alignment. Participants will complete two supervised sessions per week and perform home exercises twice daily (10 repetitions per exercise) for 6 weeks. Exercise adherence will be tracked with an exercise diary, and participants who miss the program for three consecutive days will be withdrawn from the study.
  Arms: Thoracic Stabilization Exercise Group (TSG)

SUMMARY:
This randomized controlled trial aims to compare the effects of Dynamic Neuromuscular Stabilization (DNS) exercises and thoracic stabilization exercises on thoracic erector spinae muscle strength, thoracic kyphosis angle, pain and trunk stabilization in individuals with thoracic kyphosis. Thirty participants aged 18-40 years with thoracic kyphosis will be randomly allocated to a DNS exercise group or a thoracic stabilization exercise group. Surface EMG biofeedback will be used to assess thoracic erector spinae muscle activation, while pain, thoracic kyphosis angle and trunk endurance will be evaluated using validated clinical tests. The interventions will be applied for 6 weeks, and outcomes will be assessed before and after the intervention period.

DETAILED DESCRIPTION:
Thoracic kyphosis is a frequently observed postural deviation that affects the sagittal alignment of the spine and may lead to alterations in muscular balance, impaired trunk stability, and increased biomechanical stress on the vertebral column. Postural thoracic kyphosis typically results from prolonged sedentary behaviors-such as extended computer and smartphone use-and habitual forward-flexed postures adopted during work or daily activities. Over time, inadequate thoracic extension, weakness of the thoracic erector spinae musculature, and compensatory recruitment of accessory trunk muscles may further contribute to the progression of the deformity. Although postural kyphosis is considered flexible and reversible in early stages, insufficient management may allow gradual transition toward more structural changes.

Conservative physiotherapy interventions represent the primary approach to managing postural thoracic kyphosis. These interventions traditionally include thoracic mobility exercises, strengthening of the spinal extensors, scapular stabilization strategies, and postural retraining. In recent years, neuromuscular re-education methods and biofeedback-supported interventions have become increasingly prominent, reflecting a shift toward approaches that emphasize sensorimotor control and integration of respiratory-postural synergy.

Dynamic Neuromuscular Stabilization (DNS) is a rehabilitation method grounded in developmental kinesiology principles. DNS aims to restore optimal joint stabilization and postural alignment through coordinated activation of the diaphragm, deep spinal stabilizers, and global trunk musculature. By replicating developmental postures, DNS seeks to reintegrate diaphragmatic breathing patterns and promote central stabilization strategies that influence thoracic alignment and motor control.

Thoracic stabilization exercises represent another commonly applied approach and typically include targeted thoracic extension, scapular retraction, and segmental mobilization techniques. These exercises aim to improve local muscle function of the thoracic erector spinae, enhance thoracic mobility, and promote more efficient load transfer across the spine. While both DNS and thoracic stabilization approaches have theoretical and clinical justification, direct comparative evidence regarding their short-term effects on neuromuscular activation and postural correction in adults with thoracic kyphosis remains limited.

This single-center randomized controlled trial will be conducted at Mudanya University and will include 30 adults aged 18 to 40 years with postural thoracic kyphosis confirmed through flexible ruler assessment. Participants will be randomly assigned in a 1:1 ratio to either a Dynamic Neuromuscular Stabilization intervention group or a Thoracic Stabilization Exercise group. Both intervention programs will extend over a 6-week period and will include two supervised sessions per week, complemented by home-based exercises performed twice daily. To ensure adherence, each participant will maintain an exercise diary, and individuals who fail to perform the prescribed exercises for three consecutive days will be withdrawn from the study in accordance with predefined adherence criteria.

Outcome measures will be collected at baseline and after the 6-week intervention. Surface electromyography (EMG) biofeedback will be used to assess thoracic erector spinae muscle activity. Pain intensity will be evaluated using the Visual Analog Scale (VAS). Trunk endurance and stabilization capacity will be measured using standardized plank tests and the Biering-Sørensen back endurance test. Thoracic curvature will be quantified using a flexible ruler, from which a kyphosis index will be calculated. Additional data-such as demographic characteristics, body mass index, and relevant medical history-will be recorded to contextualize findings and ensure appropriate characterization of the study population.

The primary aim of this trial is to compare the effects of DNS and thoracic stabilization exercises on thoracic erector spinae muscle activation measured via EMG. Secondary objectives include comparing the influence of both interventions on thoracic kyphosis angle, pain intensity, and trunk stabilization performance. The study is designed to provide a detailed evaluation of two physiotherapy approaches grounded in distinct theoretical frameworks, thereby offering insight into their mechanisms and potential applicability for individuals presenting with postural thoracic kyphosis. Findings will be reported separately in the Results section once data collection and analysis are completed. The present description outlines the scientific rationale and methodological approach without including results or interpretations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years.
* Presence of thoracic kyphosis based on clinical and flexible ruler assessment.
* Able to perform exercise-based interventions.
* Voluntarily agrees to participate and signs the informed consent form.
* No neurological, systemic, cardiac or orthopedic condition that would prevent safe participation in the exercise program.

Exclusion Criteria:

* Age outside the range of 18-40 years.
* Pregnancy.
* Malignancy.
* History of spinal surgery within the last year.
* Currently performing spinal or intensive core stabilization exercises.
* Visual, auditory or cognitive impairment that would interfere with cooperation during the intervention.
* Contraindications to exercise participation.
* Non-adherence to the exercise program (not performing exercises for three consecutive days).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Thoracic Kyphosis Index (Flexible Ruler Measurement) | Baseline and Week 6
  Thoracic kyphosis will be measured using a flexible ruler placed from C7 to T12 in standing posture. The curve will be transferred to paper and the kyphosis index will be calculated using the formula (H/U) × 100, where H is the height and U is the length of the curve. Higher scores indicate greater kyphosis.
  Analysis Metric:
  Change from baseline to Week 6 in kyphosis index.

SECONDARY OUTCOMES:
Thoracic Erector Spinae Muscle Activity (Surface EMG, µV) | Baseline and Week 6
  Thoracic erector spinae muscle activity will be evaluated using surface EMG biofeedback. Surface electrodes will be placed along the thoracic erector spinae musculature. Participants will perform standardized isometric contractions, and mean microvolt (µV) amplitudes will be recorded at baseline and after 6 weeks of intervention.
  Analysis Metric:
  Change from baseline to Week 6 in mean EMG amplitude (µV).
Pain Intensity - Visual Analog Scale (VAS) | Baseline and Week 6
  Pain intensity will be assessed using a 10-cm Visual Analog Scale, where 0 indicates no pain and 10 indicates worst imaginable pain. Participants will rate their pain at baseline and after 6 weeks.
  Analysis Metric:
  Change from baseline to Week 6 in VAS score.
Plank Test (Core Endurance, seconds) | Baseline and Week 6
  Core muscle endurance will be assessed using the prone plank test. Participants will maintain a standardized prone plank position supported on forearms and toes for as long as possible. Time to fatigue (seconds) will be recorded.
  Analysis Metric:
  Change from baseline to Week 6 in plank hold time (seconds).
Lateral Plank Test (Oblique Endurance, seconds) | Baseline and Week 6
  Lateral plank tests will be used to assess lateral trunk endurance. Participants will support their body on one elbow and the side of the foot, maintaining a straight alignment. Time to fatigue will be recorded separately for both sides.
  Analysis Metric:
  Change from baseline to Week 6 in side plank hold time (seconds).
Sorensen Back Extensor Endurance Test (seconds) | Baseline and Week 6
  Back extensor endurance will be evaluated using the Biering-Sørensen test. With the lower body fixed to the examination table at the level of the iliac crests, participants will maintain the upper body in a horizontal position unsupported as long as possible. Time to fatigue (seconds) will be recorded.
  Analysis Metric:
  Change from baseline to Week 6 in endurance time (seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Esra Beceni, Lecturer, Study Director — Mudanya University Vocational School , Physiotherapy Program"; Server Erdoğmuş Gülcan, PhD students, Principal Investigator — Mudanya University, Faculty of Health Sciences, Department of Physiotherapy; Ata Ekşi, Undergraduate student, Study Chair — Mudanya University, Faculty of Health Sciences, Department of Physiotherapy
Locations (1):
- Mudanya University, Bursa, Turkey (Türkiye)